CLINICAL TRIAL: NCT01141283
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study of the Efficacy and Safety of Buprenorphine Transdermal System (BTDS) in Subjects With Mod to Sev OA Pain of Hip or Knee: A 6-Month Open-label Extension Phase
Brief Title: Safety of BTDS in Subjects With Osteoarthritic (OA) Pain of Hip or Knee: A 6-Month Open-label Extension Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP3012S
Record Dates: First submitted 2010-06-02; First posted 2010-06-10 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Opioid; Transdermal
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BTDS (Experimental): Buprenorphine transdermal patch
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 5 mcg/h applied for 7-day wear
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 10 mcg/h applied for 7-day wear
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 20 mcg/h applied for 7-day wear

SUMMARY:
The purpose of the extension phase is to evaluate the long-term safety and tolerability of buprenorphine transdermal system (BTDS).

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain. Transdermal systems may offer advantages over currently indicated oral products including ease and convenience of use, improved compliance, possible reduction in patient care, and prolonged and consistent delivery of drug.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe osteoarthritic (OA) pain who completed all visits of the double-blind phase on study drug, or who discontinued study drug due to lack of therapeutic effect in the double-blind phase, but still completed all visits of the double-blind phase off study drug, are eligible to enroll in the extension phase.

Exclusion Criteria:

* Excluded from the study are subjects who ingest > 2500 mg/day acetaminophen as part of their current stable nonopioid analgesic regimen.
* Subjects requiring long-acting opioid analgesics [once- or twice-daily dosing with an every (q) 24 hour (h) or q12h drug] or transdermal fentanyl during the extension phase should be discontinued from the study.

Refer to core study for additional inclusion/exclusion information.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2003-04; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Vista Medical Research Inc., Mesa, Arizona
  - Arthrocare, Arthritis Care and Research, Phoenix, Arizona
  - Arizona Rheumatology Ctr and Phoenix Ctr for Clinical Research, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Research Facility, Tucson, Arizona
  - Advanced Pain Medicine, Bakersfield, California
  - Orange County Clinical Research, Cypress, California
  - San Diego Arthritis & Osteoporosis Medical Clinic, San Diego, California
  - Research Facility, San Diego, California
  - Research Facility, San Francisco, California
  - Research Facility, Denver, Colorado
  - Research Facility, Westminster, Colorado
  - Research Facility, Bridgeport, Connecticut
  - Research Facility, Atlantis, Florida
  - Allergy, Asthma, Arthritis & Lung, Daytona Beach, Florida
  - University Clinical Research Deland, DeLand, Florida
  - Research Facility, Jupiter, Florida
  - Coastal Medical Research, Orange City, Florida
  - Research Facility, Plantation, Florida
  - Research Facility, West Palm Beach, Florida
  - Research Facility, Marietta, Georgia
  - Research Facility, Columbus, Indiana
  - Research Facility, Evansville, Indiana
  - Primary Care Medical Center, Murray, Kentucky
  - Great Lakes Family Care, Cadillac, Michigan
  - Research Facility, Traverse City, Michigan
  - Beth Israel/Dept. of Pain, New York, New York
  - Research Facility, Winston-Salem, North Carolina
  - Research Facility, Cresson, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University Orthopedics & Sport Medicine Center, State College, Pennsylvania
  - Research Facility, West Reading, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Central Plains Clin-Brown Site, Watertown, South Dakota
  - Research Facility, Dallas, Texas
  - Research Facility, Harker Heights, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Seguin, Texas
  - Granger Medical Clinic, West Valley City, Utah
  - Hilltop Medical Center, Virginia Beach, Virginia
  - Research Facility, Bellevue, Washington
  - Internal Medicine Northwest, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28-May-2003 (first patient first visit) to 02-Jul-2004 (last patient last visit of extension phase). This study was conducted at 11 medical/research sites in the U.S.
Pre-assignment Details: All subjects meeting the protocol-specified definition of "double blind phase completer" were eligible to participate in the extension phase within 3 days. Completers were defined as those who either developed inadequate analgesia in the double-blind phase or completed all 28 days of the double-blind phase on study drug with adequate analgesia.
Groups:
- Extension Phase (BTDS 5, 10, or 20): Buprenorphine transdermal patches of BTDS 5, 10, or 20 applied for 7-day wear
Period: Overall Study
Arm/Group | Extension Phase (BTDS 5, 10, or 20)
Started | 290
Completed | 202
Not Completed | 88
Not completed — Adverse Event | 56
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 14
Not completed — Administrative | 4
Not completed — Lack of Efficacy | 10

BASELINE CHARACTERISTICS:
Arm/Group | Extension Phase (BTDS 5, 10, or 20)
Number analyzed (Participants) | 290
Age Continuous [Mean (Standard Deviation); unit: years] | 60.4 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197
  Male | 93

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Safety was assessed using reports of adverse events, clinical laboratory results, findings from physical examinations, and vital sign measurements.
Time Frame: 6 months.
Population: The extension safety population consisted of all subjects who were exposed to BTDS and had at least 1 safety assessment during extension phase.
Measure: Number; unit: participants
Arm/Group | Extension Phase (BTDS 5, 10, or 20)
Number analyzed (Participants) | 290
participants
  Deaths | 0 (0)
  Serious Adverse Events | 6
  Adverse Events 4.5% | 202

ADVERSE EVENTS:
Time Frame: Adverse events ongoing at study completion must be followed until resolution or for 30 days after the last dose of study drug, whichever comes first. SAEs must be followed until the event resolves or the event or sequelae stabilize.
Description: Adverse events were obtained through spontaneous reports and subject interview.
Arm/Group | Extension Phase (BTDS 5, 10, or 20)
Serious Adverse Events (participants affected / at risk) | 6/290
Other Adverse Events (participants affected / at risk) | 202/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extension Phase (BTDS 5, 10, or 20) (N=290)
Chest pain (General disorders) | 1 (1) — Systematic and nonsystematic assessments.
Chest pain atypical (General disorders) | 1 (1) — Systematic and nonsystematic assessments.
Left foot osteomyelitis (Infections and infestations) | 1 (1) — Systematic and nonsystematic assessments.
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) — Systematic and nonsystematic assessments.
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) — Systematic and nonsystematic assessments.
Exacerbation of osteoarthritis (OA) in the right knee (Musculoskeletal and connective tissue disorders) | 1 (1) — Systematic and nonsystematic assessments.
Transient ischemic attack (Nervous system disorders) | 1 (1) — Systematic and nonsystematic assessments.
Dysarthria (Nervous system disorders) | 1 (1) — Systematic and nonsystematic assessments.
Left lateral intraventricular hemorrhage (Nervous system disorders) | 1 (1) — Systematic and nonsystematic assessments.
Seizure (Nervous system disorders) | 1 (1) — Systematic and nonsystematic assessments.
Syncopal episode (Nervous system disorders) | 1 (1) — Systematic and nonsystematic assessments.
Diabetic ulceration left foot (Skin and subcutaneous tissue disorders) | 1 (1) — Systematic and nonsystematic assessments.
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Extension Phase (BTDS 5, 10, or 20) (N=290)
Nausea (Gastrointestinal disorders) | 38 — Systematic and nonsystematic assessments.
Constipation (Gastrointestinal disorders) | 37 — Systematic and nonsystematic assessments.
Vomiting NOS (Gastrointestinal disorders) | 17 — Systematic and nonsystematic assessments.
Application site pruritus (General disorders) | 36 — Systematic and nonsystematic assessments.
Application site rash (General disorders) | 39 — Systematic and nonsystematic assessments.
Application site erythema (General disorders) | 39 — Systematic and nonsystematic assessments.
Application site irritation (General disorders) | 19 — Systematic and nonsystematic assessments.
Upper respiratory tract infection NOS (Infections and infestations) | 17 — Systematic and nonsystematic assessments.
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 — Systematic and nonsystematic assessments.
Back pain (Musculoskeletal and connective tissue disorders) | 35 — Systematic and nonsystematic assessments.
Pain in limb (Musculoskeletal and connective tissue disorders) | 22 — Systematic and nonsystematic assessments.
Headache (Nervous system disorders) | 66 — Systematic and nonsystematic assessments.
Somnolence (Nervous system disorders) | 14 — Systematic and nonsystematic assessments.
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 19 — Systematic and nonsystematic assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days